CLINICAL TRIAL: NCT01536197
Title: Effect of Bariatric Surgery-induced Weight Loss on Taste Perception
Brief Title: Taste Perception Pre and Post Bariatric Surgery
Acronym: RBtaste
Status: Completed | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: 09-0175B
Record Dates: First submitted 2012-02-09; First posted 2012-02-20 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-11

CONDITIONS: Morbid Obesity
Keywords: obesity; gastric bypass; gastric banding; sleeve gastrectomy; weight loss; taste perception
MeSH Terms: conditions — Obesity, Morbid; Obesity; Weight Loss | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tongue tissue
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Gastric Bypass: morbidly obese subjects undergoing gastric bypass surgery
  Interventions: Procedure: Gastric bypass
- Gastric banding: morbidly obese subjects undergoing laparoscopic gastric banding surgery
  Interventions: Procedure: Gastric banding
- Sleeve gastrectomy: morbidly obese subjects undergoing sleeve gastrectomy surgery
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Gastric bypass — Roux-en-Y gastric bypass
  Groups: Gastric Bypass
Procedure: Gastric banding — Laparoscopic adjustable gastric banding
  Groups: Gastric banding
Procedure: Sleeve gastrectomy — Sleeve gastrectomy surgery
  Groups: Sleeve gastrectomy

SUMMARY:
The investigators wish to study the effects of three forms of bariatric surgery, gastric bypass lap banding, and sleeve gastrectomy. The surgery is not part of the clinical trial. If your insurance does not cover the procedure, then the patient is responsible for payment of the surgical process. The investigators are doing pre and post surgery testing to provide a better understanding of the effect of bariatric surgery-induced weight-loss on taste perception.

DETAILED DESCRIPTION:
Bariatric surgery is the most effective weight loss therapy for obesity. However, the mechanisms responsible for decreased food intake are incompletely understood. One possible mechanism that could account for decreased food intake is changes in taste perception. Therefore, the primary goal of this proposal is to provide a better understanding of the effects of bariatric surgery-induced weight-loss on taste perception.

ELIGIBILITY:
Inclusion Criteria:

* BMI >=35 kg/m²
* on stable dose of medication for at least 4 weeks before the pre-surgery studies
* women

Exclusion Criteria:

* smokes > 7 cigarettes per day
* previous malabsorptive or restrictive intestinal surgery
* pregnant or breastfeeding
* recent history of neoplasia (< 5 years ago)
* have malabsorptive syndromes and inflammatory intestinal disease
* diabetes mellitus
* show signs of oral disease or xerostomia (i.e. dry mouth)
* history of chronic rhinitis
* on medication that might affect taste
* severe organ disfunction

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 41 morbidly obese (BMI>=35 kg/m²) subjects scheduled for bariatric surgical procedures will participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Klein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gastric Bypass | Gastric Banding
Started | 23 | 10
Completed | 23 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gastric Bypass | Gastric Banding | Total
Number analyzed (Participants) | 23 | 10 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (9.6) | 46.8 (13.9) | 43.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 10 | 30
  Male | 3 | 0 | 3
Body weight before surgery [Mean (Standard Deviation); unit: Kg] | 129.8 (26.1) | 127.1 (31.0) | 128.7 (27.2)

OUTCOME MEASURES:

1. Primary Outcome: Changes on Taste Detection Thresholds After Bariatric Surgery-induced Weight Loss (Roux-en-Y Gastric Bypass and Laparoscopic Adjustable Banding).
Description: -Taste detection thresholds measures the lowest concentration of a tastant that can be detected (mili molar amounts).
Time Frame: we will measure the above outcomes before surgery and at 20% weight loss post surgery, which on average we expect will occur around 3 months post-surgery
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Gastric Bypass | Gastric Banding
Number analyzed (Participants) | 23 | 10
mmol/L
  Sucrose taste detection threshold before surgery | 7.5 [2.4 to 12.6] | 8.1 [6.5 to 11.5]
  Sucrose taste detection threshold after surgery | 6.5 [4.6 to 8.4] | 7.5 [4.9 to 13.4]
Statistical Analysis 1: Comparison: Gastric Bypass vs Gastric Banding; Test type: Superiority or Other; p = 0.19, ANOVA; Two-way ANOVAs with group (gastric bypass and lap banding) as the between-subjects factor and time (before after surgery)

2. Secondary Outcome: Changes on Emotional, External and Restricted Eating Behavior and Food Craving After Bariatric Surgery-induced Weight Loss (Roux-en-Y Gastric Bypass and Laparoscopic Adjustable Gastric Banding).
Description: -Eating behavior will be measured with validated questionnaires including among others the Dutch Eating Behavior Questionnaire (DEBQ) and the Food Craving Inventory (FCI). The DEBQ measures three common psychological dimensions of eating behavior: 1) emotional eating , 2) external eating (an inclination to eat in response to external food cues such as the smell and taste of food), and 3) restrained eating (an inclination to consciously restrict food intake to control body weight). The FCI is a validated measure of the frequency of overall food cravings as well as cravings for specific types of foods (high fats, sweets, carbohydrates/ starches, and fast-food fats) during the past month. For the DEBQ and the FCI, subjects score their answers by using a 5-point Likert scale (1=never, 5=very often/always).Therefore, lower numbers means having less frequent food cravings (for FCI), or engaging less frequently in the particular type of eating behavior (for DEBQ).
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Gastric Bypass | Gastric Banding
Number analyzed (Participants) | 23 | 10
units on a scale
  Cravings for sweets before surgery | 2.3 (0.8) | 2.7 (0.7)
  Cravings for sweets after surgery | 1.6 (0.6) | 2.3 (0.5)
  Cravings for fast food before surgery | 2.9 (0.7) | 2.6 (0.8)
  Cravings for fast food after surgery | 2.2 (0.6) | 2.2 (0.5)
  Cravings for high fat food before surgery | 2.2 (0.7) | 2.0 (0.8)
  Cravings for high fat food after surgery | 1.8 (0.6) | 1.9 (0.7)
  Cravings for starchy food before surgery | 2.2 (0.8) | 2.2 (0.5)
  Cravings for starchy food after surgery | 1.9 (0.7) | 1.9 (0.6)
  Restrained eating before surgery | 2.9 (0.6) | 2.8 (0.5)
  Restrained eating after surgery | 3.0 (0.7) | 3.4 (1)
  Emotional eating before surgery | 2.6 (0.9) | 3.2 (1.0)
  Emotional eating after surgery | 1.8 (0.7) | 2.3 (1.0)
  External eating before surgery | 3.0 (0.5) | 3.4 (0.5)
  External eating after surgery | 2.2 (0.5) | 2.4 (0.6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Gastric Bypass | Gastric Banding
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/10
Other Adverse Events (participants affected / at risk) | 0/23 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No